CLINICAL TRIAL: NCT00764881
Title: Multi-center, Double-blind, Randomized Study to Investigate the Impact of a Sequential Oral Contraceptive Containing Estradiol Valerate and Dienogest (SH T00658ID) Compared to a Monophasic Contraceptive Containing Ethinylestradiol and Levonorgestrel (Microgynon) Over 6 Treatment Cycles on Alleviating Complaints of Reduced Libido in Women With Acquired Female Sexual Dysfunction (FSD) Associated With Oral Contraceptive Use
Brief Title: Effects of SH T00658ID on Libido
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91548; 2008-002263-13 (EudraCT Number); 310785 (Other: Company Internal)
Record Dates: First submitted 2008-10-01; First posted 2008-10-02 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Contraception; Libido
Keywords: Oral contraceptive; Sexual dysfunction; Libido
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — ethinyl estradiol, levonorgestrel drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) (Experimental): Daily oral administration of one capsule BAY86-5027 [estradiol valerate (EV) / dienogest (DNG)] for 28 days per cycle in the sequential 4-phasic regimen for 6 treatment cycles.
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658ID)
- EE/LNG (Microgynon) + Placebo (Active Comparator): Daily oral administration of one capsule ethinylestradiol (EE) / levonorgestrel (LNG) for 21 days, followed by 1 capsule placebo for 7 days (28 days total per cycle) for 6 treatment cycles.
  Interventions: Drug: Microgynon; Drug: Placebo

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658ID) — Estradiol valerate (EV) and dienogest (DNG). Sequential 4-phasic regimen. Daily oral administration of one encapsulated SH T00658ID for 28 days per cycle, for 6 treatment cycles: Days 1-2, 3.0 mg EV; Days 3-7, 2.0 mg EV+2.0 mg DNG; Days 8-24, 2.0 mg EV+3.0 mg DNG; Days 25-26, 1.0 mg EV; Days 27-28, placebo, encapsulated for blinding purpose
  Arms: EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID)
Drug: Microgynon — Days 1 to 21: daily oral administration of one encapsulated Microgynon tablet; 0.03 mg ethinylestradiol (EE) + 0.15 mg levonorgestrel (LNG). Six 28-day treatment cycles.
  Arms: EE/LNG (Microgynon) + Placebo
Drug: Placebo — Days 22 to 28: daily oral administration of one encapsulated placebo tablet. Six 28-day treatment cycles.
  Arms: EE/LNG (Microgynon) + Placebo

SUMMARY:
The aim of the study is to investigate whether women on oral contraceptives (OCs) suffering from acquired OC-associated female sexual dysfunction (FSD) for at least 3 months but no longer than one year will express the same level of sexual distress when taking SH T00658ID compared to Microgynon, the usual OC prescribed for women with OC-associated FSD.

ELIGIBILITY:
Inclusion Criteria:

* OC-associated female sexual dysfunction (FSD) for at least 3 months but no longer than one year and willingness to continue OC use but to switch to SH T00658ID or Microgynon
* Combined score of the sexual desire and arousal domains of the FSFI questionnaire of 18 or below at screening and baseline

Exclusion Criteria:

* Contraindications for oral contraceptive use, for example but not limited to: presence or history of venous or arterial thrombotic / thromboembolic events, hypertension, presence or history of severe hepatic disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 217 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (32):
- Australia (6):
  - Sydney Centre for Reproductive Health Reseach, Ashfield, New South Wales
  - Royal Hospital for Women, Sydney, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Prahran, Victoria
  - Queen Elizabeth II Medical Centre, Nedlands, Western Australia
  - King Edward Memorial Hospital, Subiaco, Western Australia
- Austria (7):
  - Ordination Dr. Schmidl-Amann, Sankt Pölten, Lower Austria
  - Ordination Dr.Hohlweg, Graz, Styria
  - Ordination Dr. Schaffer, Graz, Styria
  - Clin Pharm International GmbH Studienzentrum Wien, Vienna, Vienna
  - Dr. Brigitte Wiesenthal, Vienna
  - Dr. Wolfgang Bartl, Vienna
  - Dr. Walter Paulik, Zeltweg
- Belgium (3):
  - Hôpital Erasme/Erasmus Ziekenhuis, Bruxelles - Brussel
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Germany (4):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Praxis Dr. A. Schwenkhagen-Stodieck, Hamburg, Hamburg
  - Universitätsklinikum Aachen, Aachen, North Rhine-Westphalia
  - Frauenarztpraxis Dr. Bernd Pittner, Leipzig, Saxony
- Italy (4):
  - A.O.U. di Cagliari, Monserrato, Cagliari
  - A.O.U. Policlinico - Vittorio Emanuele, Catania
  - IRCCS Fondazione Maugeri - Montescano (Pavia), Pavia
  - A.O.U. Pisana, Pisa
- Spain (5):
  - Centro de Planificacion Familiar Alicante 3, Alicante, Alicante
  - USP Institut Universitari Dexeus, Barcelona, Barcelona
  - Diatros Gava- Centre Assistencial Ntra. Sra. de Burgues, Gavà, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Instituto Palacios de Salud y Medicina de la Mujer, Madrid
- Thailand (3):
  - Chulalongkorn Hospital, Bangkok
  - Ramathibodhi Hospital, Bangkok
  - Siriraj Hospital, Mahidol, Bangkok

REFERENCES:
- [Derived] Davis SR, Bitzer J, Giraldi A, Palacios S, Parke S, Serrani M, Mellinger U, Nappi RE. Change to either a nonandrogenic or androgenic progestin-containing oral contraceptive preparation is associated with improved sexual function in women with oral contraceptive-associated sexual dysfunction. J Sex Med. 2013 Dec;10(12):3069-79. doi: 10.1111/jsm.12310. Epub 2013 Sep 12. PMID 24034466
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The date of first subject was 29 Jan 2009. The date of last subject was 20 Jul 2010.
Pre-assignment Details: Of 276 participants screened, 29 failed Screening, and 217 were randomized 1:1, of which 1 never received treatment, 3 had no observations, and 213 were treated (EV/DNG=106; EE/LNG=107).
Period: Overall Study
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Started | 108 | 109
Subjects Received Treatment | 106 (Full Analysis Set (FAS)) | 107 (Full Analysis Set (FAS))
Completed | 92 | 99
Not Completed | 16 | 10
Not completed — Adverse Event | 5 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Protocol Violation | 2 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Noncompliant | 1 | 0
Not completed — Accidentally discontinued study drug | 1 | 0
Not completed — Wished to become pregnant | 1 | 0
Not completed — Carcinoma detected | 1 | 0
Not completed — Possibly noncompliant (study drug) | 0 | 2
Not completed — no treatment or no observation | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo | Total
Number analyzed (Participants) | 106 | 107 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (7.0) | 30.2 (7.8) | 30.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 107 | 213
  Male | 0 | 0 | 0
Ethnic group [Number; unit: participants]
  Caucasian | 90 | 92 | 182
  Hispanic | 0 | 1 | 1
  Asian | 16 | 13 | 29
  Other | 0 | 1 | 1
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 22.8 (3.2) | 22.7 (2.9) | 22.8 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Cycle 6 in the Total of Questions 1 to 6 of the Female Sexual Function Index (FSFI) - Full Analysis Set (FAS)
Description: Change from Baseline FSFI domains in desire and arousal component scores at Cycle 6. The change in score ranges from -28 (worst) to 28 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
scores on a scale | 6.45 (5.33) | 5.98 (6.22)

2. Primary Outcome: Change From Baseline to Cycle 6 in the Total of Questions 1 to 6 of the Female Sexual Function Index (FSFI) - Per Protocol Set (PPS)
Description: as for outcome 1
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: Per Protocol Set (PPS) includes those participants of the FAS without major protocol deviations affecting the primary variables
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 92 | 95
scores on a scale | 6.43 (5.36) | 6.37 (5.86)

3. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Desire) at Baseline
Description: Sum of questions 1 and 2 on sexual desire on the FSFI Questionnaire at Baseline. The normalized score for those 2 questions ranges from 1.2 (worst) to 6 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
scores on a scale | 2.51 (0.72) | 2.39 (0.74)

4. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Desire) at Cycle 6
Description: Sum of questions 1 and 2 on sexual desire on the FSFI Questionnaire at Cycle 6. The normalized score for those 2 questions ranges from 1.2 (worst) to 6 (best).
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
scores on a scale | 3.53 (0.95) | 3.52 (0.89)

5. Secondary Outcome: Mean Change From Baseline to Cycle 6 in FSFI Domain Score (Desire)
Description: Mean change from Baseline to Cycle 6 in the sum of questions 1 and 2 on sexual desire on the FSFI Questionnaire. The change in the normalized score for those 2 questions ranges from -4.8 (worst) to 4.8 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
scores on a scale | 1.02 (0.98) | 1.11 (1.02)

6. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Arousal) at Baseline
Description: Sum of questions 3 to 6 on sexual arousal on the FSFI Questionnaire at Baseline. The normalized score for those 4 questions ranges from 0 (worst) to 6 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
scores on a scale | 2.65 (0.94) | 2.77 (0.83)

7. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Arousal) at Cycle 6
Description: Sum of questions 3 to 6 on sexual arousal on FSFI Questionnaire at Cycle 6. The normalized score for those 4 questions ranges from 0 (worst) to 6 (best).
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
scores on a scale | 4.03 (1.23) | 4.05 (1.35)

8. Secondary Outcome: Mean Change From Baseline to Cycle 6 in FSFI Domain Score (Arousal)
Description: Mean change from Baseline to Cycle 6 in the sum of questions 3 to 6 on sexual arousal on the FSFI Questionnaire. The change in the normalized score for those 4 questions ranges from -6 (worst) to 6 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
scores on a scale | 1.43 (1.25) | 1.24 (1.53)

9. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Lubrication) at Baseline
Description: Sum of questions 7 to 10 on lubrication on the FSFI Questionnaire at Baseline. The normalized score for those 4 questions ranges from 0 (worst) to 6 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 3.56 (1.44) | 3.73 (1.14)

10. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Lubrication) at Cycle 6
Description: Sum of questions 7 to 10 on lubrication on the FSFI Questionnaire at Cycle 6. The normalized score for those 4 questions ranges from 0 (worst) to 6 (best).
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
scores on a scale | 4.90 (1.18) | 4.81 (1.46)

11. Secondary Outcome: Mean Change From Baseline to Cycle 6 in FSFI Domain Score (Lubrication)
Description: Mean change from Baseline at Cycle 6 in the sum of questions 7 to 10 on the FSFI Questionnaire. The change in the normalized score for those 4 questions ranges from -6 (worst) to 6 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 1.36 (1.53) | 1.04 (1.91)

12. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Orgasm) at Baseline
Description: Sum of questions 11 to 13 on orgasm on FSFI Questionnaire at Baseline. The normalized score for those 3 questions ranges from 0 (worst) to 6 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 2.97 (1.41) | 2.93 (1.24)

13. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Orgasm) at Cycle 6
Description: Sum of questions 11 to 13 on orgasm on the FSFI Questionnaire at Cycle 6. The normalized score for those 3 questions ranges from 0 (worst) to 6 (best).
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 4.22 (1.52) | 4.05 (1.49)

14. Secondary Outcome: Mean Change From Baseline to Cycle 6 in FSFI Domain Score (Orgasm)
Description: Mean change from Baseline to Cycle 6 in the sum of questions 11 to 13 on orgasm on the FSFI Questionnaire. The change in the normalized score for those 3 questions ranges from -6 (worst) to 6 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 1.26 (1.52) | 1.06 (1.65)

15. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Satisfaction) at Baseline
Description: Sum of Questions 14 to 16 on satisfaction on the FSFI Questionnaire at Baseline. The normalized score for those 3 questions ranges from 0.8 (worst) to 6 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 3.16 (1.06) | 3.20 (0.78)

16. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Satisfaction) at Cycle 6
Description: Sum of questions 14 to 16 on satisfaction on the FSFI Questionnaire at Cycle 6. The normalized score for those 3 questions ranges from 0.8 (worst) to 6 (best).
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 4.19 (1.13) | 4.26 (1.10)

17. Secondary Outcome: Mean Change From Baseline to Cycle 6 in FSFI Domain Score (Satisfaction)
Description: Mean change from Baseline to Cycle 6 in the sum of questions 14 to 16 on satisfaction on the FSFI Questionnaire. The change in the normalized score for those 3 questions ranges from -5.2 (worst) to 5.2 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 1.03 (1.24) | 1.03 (1.20)

18. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Pain) at Baseline.
Description: Sum of questions 17 to 19 on pain on the FSFI Questionnaire at Baseline. The normalized score for those 3 questions ranges from 0 (worst) to 6 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 4.34 (1.78) | 4.74 (1.52)

19. Secondary Outcome: The Mean Absolute Values of FSFI Domain Score (Pain) at Cycle 6
Description: Sum of questions 17 to 19 on pain on the FSFI Questionnaire at Cycle 6. The normalized score for those 3 questions ranges from 0 (worst) to 6 (best).
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 5.04 (1.53) | 5.01 (1.55)

20. Secondary Outcome: Mean Change From Baseline to Cycle 6 in FSFI Domain Score (Pain)
Description: Mean change from Baseline to Cycle 6 in the sum of questions 17 to 19 on pain on the FSFI Questionnaire. The change in the normalized score for those 3 questions ranges from -6 (worst) to 6 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 0.69 (1.83) | 0.22 (1.89)

21. Secondary Outcome: The Mean Absolute Values of FSFI Total Score at Baseline
Description: The normalized FSFI total score was the weighted sum of the domain scores covering a range from 2 (worst) to 36 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
scores on a scale | 19.2 (5.6) | 19.8 (4.8)

22. Secondary Outcome: The Mean Absolute Values of FSFI Total Score at Cycle 6
Description: The normalized FSFI total score was the weighted sum of the domain scores covering a range from 2 (worst) to 36 (best).
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 25.8 (6.5) | 25.7 (6.8)

23. Secondary Outcome: Mean Change From Baseline to Cycle 6 in FSFI Total Score
Description: The change in the normalized FSFI total score ranges from -34 (worst) to 34 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Scores on a scale | 6.7 (6.9) | 5.7 (7.8)

24. Secondary Outcome: The Mean Absolute Values of Female Sexual Distress Scale (FSDS-R) Total Score at Baseline
Description: Validated, 13-item scale (0=never to 4=always) that assesses subjective distress associated with sexual dysfunction in women. A decrease in the total score=decrease in frequency of the subjective distress symptom. The total score ranges from 0 (worst) to 52 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 25.6 (10.6) | 27.5 (10.2)

25. Secondary Outcome: The Mean Absolute Values of Female Sexual Distress Scale (FSDS-R) Total Score at Cycle 6
Description: as for outcome 24
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 14.8 (10.2) | 17.6 (11.4)

26. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Female Sexual Distress Scale (FSDS-R) Total Score
Description: Change from Baseline to Cycle 6 in the validated, 13-item scale (0=never to 4=always) that assesses subjective distress associated with sexual dysfunction in women. A decrease in the total score=decrease in frequency of the subjective distress symptom. The change in total score ranges from -52 (best) to 52 (worst).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | -10.0 (10.4) | -9.6 (10.5)

27. Secondary Outcome: The Mean Absolute Values of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) (Short Version) Total Score at Baseline
Description: Q-LES-Q (short version - 16 items) assessed at Baseline the degree of enjoyment and satisfaction during the past week taking everything into consideration on a 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 69.76 (10.85) | 68.47 (11.98)

28. Secondary Outcome: The Mean Absolute Values of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) (Short Version) Total Score at Cycle 6
Description: Q-LES-Q (short version - 16 items) assessed at Cycle 6 the degree of enjoyment and satisfaction during the past week taking everything into consideration on a 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best).
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 71.63 (11.72) | 72.48 (10.57)

29. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q) (Short Version) Total Score
Description: Change from Baseline to Cycle 6 in the overall enjoyment and satisfaction experienced during the past week as scored on the QLES-Q (short version - 16 items). 1-5 scale (very poor, poor, fair, good, very good). The normalized score ranges from 0 (worst) to 100 (best). The change in the normalized score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 2.60 (11.26) | 4.12 (10.71)

30. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) Global Score at Baseline
Description: The PGWBI measured at Baseline self-representations over the past 4 weeks of intrapersonal affective or emotional states reflecting a sense of subjective well-being or distress. The response format used a 6-grade Likert scale and the range of PGWBI scores were normalized from 0 to 100. The higher the score, the better the well-being of the participant
Time Frame: At Baseline
Population: All participants in FAS with assessment for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 105 | 107
Scores on a scale | 67.75 (6.78) | 67.98 (7.36)

31. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) Global Score at Cycle 6
Description: The PGWBI measured at Cycle 6 self-representations over the past 4 weeks of intrapersonal affective or emotional states reflecting a sense of subjective well-being or distress. The response format used a 6-grade Likert scale and the range of PGWBI scores were normalized from 0 to 100. The higher the score, the better the well-being of the participant
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 69.20 (8.32) | 69.86 (6.95)

32. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Psychological General Well-Being Index (PGWBI) Global Score
Description: Change from Baseline to Cycle 6 in the PGWBI Questionnaire's assessment of the participant's overall sense of well-being or distress. The response format used a 6-grade Likert scale and the change in the normalized PGWBI global score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 1.93 (8.11) | 1.90 (7.23)

33. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Anxiety at Baseline
Description: Anxiety is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the range of PGWBI scores were normalized from 0 to 100. The higher the score, the better the wellbeing of the participant.
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 70.3 (15.7) | 71.5 (16.1)

34. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Anxiety at Cycle 6
Description: as for outcome 33
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 74.8 (16.0) | 74.1 (15.6)

35. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Psychological General Well-Being Index (PGWBI) - Anxiety
Description: Anxiety is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the change in the normalized PGWBI - Anxiety score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 4.9 (14.9) | 2.6 (15.4)

36. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Depressed Mood at Baseline
Description: Depressed mood is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the range of PGWBI scores were normalized from 0 to 100. The higher the score, the better the wellbeing of the participant.
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 86.20 (11.38) | 85.79 (12.16)

37. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Depressed Mood at Cycle 6
Description: as for outcome 36
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 87.24 (13.15) | 89.94 (9.61)

38. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Psychological General Well-Being Index (PGWBI) - Depressed Mood
Description: Depressed mood is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the change in the normalized PGWBI - depressed mood score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 1.75 (13.17) | 4.25 (11.38)

39. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Positive Well-being at Baseline
Description: Positive well-being is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the range of PGWBI scores were normalized from 0 to 100. The higher the score, the better the wellbeing of the participant.
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 47.88 (9.05) | 48.46 (6.53)

40. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Positive Well-being at Cycle 6
Description: as for outcome 39
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 49.41 (6.63) | 49.26 (6.23)

41. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Psychological General Well-Being Index (PGWBI) - Positive Well-being
Description: Positive well-being is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the change in the normalized PGWBI - positive well-being score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 0.91 (9.81) | 0.98 (7.55)

42. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Self-control at Baseline
Description: Self-control is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the range of PGWBI scores were normalized from 0 to 100. The higher the score, the better the wellbeing of the participant.
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 66.40 (9.35) | 66.66 (8.36)

43. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Self-control at Cycle 6
Description: as for outcome 42
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 66.95 (9.53) | 67.18 (8.33)

44. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Psychological General Well-Being Index (PGWBI) - Self-control
Description: Self-control is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the change in the normalized PGWBI - self-control score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 0.02 (12.21) | 0.71 (9.84)

45. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - General Health at Baseline
Description: General health is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the range of PGWBI scores were normalized from 0 to 100. The higher the score, the better the wellbeing of the participant.
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 79.12 (14.75) | 81.00 (13.74)

46. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - General Health at Cycle 6
Description: as for outcome 45
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 80.22 (13.95) | 81.17 (13.31)

47. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Psychological General Well-Being Index (PGWBI) - General Health
Description: General health is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale the change in the normalized PGWBI general health score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 0.93 (15.57) | -0.15 (14.14)

48. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Vitality at Baseline
Description: Vitality is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the range of PGWBI scores were normalized from 0 to 100. The higher the score, the better the wellbeing of the participant.
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 60.27 (10.81) | 60.93 (9.01)

49. Secondary Outcome: The Mean Absolute Values of Psychological General Well-Being Index (PGWBI) - Vitality at Cycle 6
Description: as for outcome 48
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 61.83 (9.46) | 63.58 (8.31)

50. Secondary Outcome: Mean Change From Baseline to Cycle 6 in Psychological General Well-Being Index (PGWBI) - Vitality
Description: Vitality is 1 of 6 dimensions of the PGWBI self-report questionnaire used to measure the subjective well-being or distress of the participant. The response format used a 6-grade Likert scale and the change in the normalized PGWBI - vitality score ranges from -100 (worst) to 100 (best).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 1.42 (10.11) | 2.65 (10.07)

51. Secondary Outcome: Percentage of Participants With Improvement in the Investigator's Assessment in Clinical Global Impression (CGI) at Cycle 6
Description: CGI is used to collect information regarding the subject's total clinical experience. The assessment scale ranges from 0 to 7: (0=not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse). The scale of 1, 2, and 3 were categorized as improvement.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Percentage of participants | 68.1 | 70.5

52. Secondary Outcome: Percentage of Participants With Improvement in Participant's Assessment in Clinical Global Impression (CGI) at Cycle 6
Description: In 1 section of the CGI the subject rates their total improvement and rate of satisfaction with sexuality during treatment. The assessment scale ranges from 0 to 7: (0=not assessed; 1=very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse). The scale of 1, 2, and 3 were categorized as improvement.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Percentage of participants | 70.3 | 62.7

53. Secondary Outcome: Vaginal Effects Evaluated by Vaginal pH at Cycle 6
Description: Vaginal pH (0 to 6) measured by subject using a pH indicator dipstick
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Proportion of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 102
Proportion of participants
  Vaginal pH < 4.0 | 0.053 | 0.039
  Vaginal pH 4.0 - 4.4 | 0.298 | 0.294
  Vaginal pH 4.5 - 5.0 | 0.521 | 0.637
  Vaginal pH > 5.0 | 0.117 | 0.029

54. Secondary Outcome: Vaginal Effects Evaluated by the Mean Absolute Values of Atrophy Symptom Questionnaire (ASQ) at Baseline
Description: ASQ consists of 5 items which define the status of the vagina. The response format uses a 4-point scale from 0 (none) to 3 (severe).
Time Frame: At Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 106 | 107
Scores on a scale | 0.54 (0.55) | 0.47 (0.48)

55. Secondary Outcome: Vaginal Effects Evaluated by the Mean Absolute Values of Atrophy Symptom Questionnaire (ASQ) at Cycle 6
Description: as for outcome 54
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 0.27 (0.40) | 0.25 (0.36)

56. Secondary Outcome: Vaginal Effects Evaluated by the Mean Change From Baseline to Cycle 6 in Atrophy Symptom Questionnaire (ASQ)
Description: ASQ consists of 5 items which define the status of the vagina. The response format uses a 4-point scale from 0 (none) to 3 (severe). The change in average score ranges from -3 (best) to 3 (worst).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | -0.27 (0.50) | -0.18 (0.38)

57. Secondary Outcome: Vaginal Effects Evaluated by the Mean Absolute Values of Vaginal Health Assessment (VHA) at Baseline
Description: The VHA, performed by the Investigator during gynecological exam, is the average of 5 individual scores related to composition and appearance of the vagina (secretions, epithelial integrity, epithelial surface thickness, color, and pH) scored from 0 (no atrophy or pH<4) to 3 (severe or pH5).
Time Frame: At Baseline
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 105 | 107
Scores on a scale | 0.33 (0.14) | 0.38 (0.26)

58. Secondary Outcome: Vaginal Effects Evaluated by the Mean Absolute Values of Vaginal Health Assessment (VHA) at Cycle 6
Description: as for outcome 57
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 93 | 102
Scores on a scale | 0.34 (0.15) | 0.31 (0.12)

59. Secondary Outcome: Vaginal Effects Evaluated by the Mean Change From Baseline to Cycle 6 in Vaginal Health Assessment (VHA)
Description: The VHA, performed by the Investigator during gynecological exam, is the average of 5 individual scores related to composition and appearance of the vagina (secretions, epithelial integrity, epithelial surface thickness, color, and pH) scored from 0 (no atrophy or pH<4) to 3 (severe or pH5). The change in average score ranges from -3 (best) to 3 (worst).
Time Frame: Baseline up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 92 | 102
Scores on a scale | 0.01 (0.18) | -0.06 (0.27)

60. Secondary Outcome: Number of Bleeding / Spotting Days in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to 90 during study treatment and includes the initial bleeding episode that triggered the first intake of study medication, meaning that the first treatment cycle includes 2 bleeding episodes.
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 99
Days | 16.3 (10.1) | 15.3 (5.6)

61. Secondary Outcome: Number of Bleeding / Spotting Days in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to 180 during study treatment
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 68 | 75
Days | 12.2 (8.2) | 12.6 (5.4)

62. Secondary Outcome: Number of Bleeding / Spotting Episodes in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to Day 90 during study treatment and includes the initial bleeding episode that triggered the first intake of study medication, meaning that the fist treatment cycle includes 2 bleeding episodes
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 99
episodes | 3.5 (1.5) | 3.3 (1.3)

63. Secondary Outcome: Number of Bleeding / Spotting Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 68 | 75
episodes | 3.0 (1.6) | 3.1 (0.7)

64. Secondary Outcome: Mean Length of Bleeding / Spotting Episodes in Reference Period 1
Description: Reference Period 1 is defined as Day 1 to Day 90 during study treatment and includes the initial bleeding episode that triggered the first intake of study medication, meaning that the first treatment cycle includes 2 bleeding episodes
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 90 | 99
Days | 4.47 (2.44) | 4.42 (1.36)

65. Secondary Outcome: Mean Length of Bleeding / Spotting Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 61 | 75
Days | 4.13 (2.09) | 4.03 (1.17)

66. Secondary Outcome: Maximum Length of Bleeding / Spotting Episodes in Reference Period 1
Description: as for outcome 64
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 90 | 99
Days | 6.6 (4.7) | 5.6 (2.6)

67. Secondary Outcome: Maximum Length of Bleeding / Spotting Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 61 | 75
Days | 5.3 (2.9) | 4.7 (1.6)

68. Secondary Outcome: Difference in Duration Between Longest and Shortest Bleeding / Spotting Episodes in Reference Period 1
Description: as for outcome 64
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 90 | 99
Days | 3.8 (4.5) | 2.2 (2.7)

69. Secondary Outcome: Difference in Duration Between Longest and Shortest Bleeding / Spotting Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 61 | 75
Days | 2.3 (2.4) | 1.3 (1.5)

70. Secondary Outcome: Number of Spotting Only Days in Reference Period 1
Description: as for outcome 64
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 99
Days | 7.6 (7.8) | 3.8 (3.9)

71. Secondary Outcome: Number of Spotting Only Days in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 68 | 75
Days | 6.1 (6.0) | 3.3 (4.7)

72. Secondary Outcome: Number of Spotting Only Episodes in Reference Period 1
Description: as for outcome 64
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 94 | 99
episodes | 1.1 (1.4) | 0.4 (1.1)

73. Secondary Outcome: Number of Spotting Only Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 68 | 75
episodes | 1.1 (1.5) | 0.4 (1.1)

74. Secondary Outcome: Mean Length of Spotting-only Episodes in Reference Period 1
Description: as for outcome 64
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 50 | 22
Days | 3.38 (3.43) | 2.79 (1.77)

75. Secondary Outcome: Mean Length of Spotting-only Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 33 | 16
Days | 3.18 (2.26) | 3.23 (2.46)

76. Secondary Outcome: Maximum Length of Spotting-only Episodes in Reference Period 1
Description: as for outcome 64
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 50 | 22
Days | 3.9 (3.5) | 3.3 (2.4)

77. Secondary Outcome: Maximum Length of Spotting-only Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 33 | 16
Days | 3.9 (2.8) | 3.7 (2.9)

78. Secondary Outcome: Difference in Duration Between Longest and Shortest Spotting-only Episodes in Reference Period 1
Description: as for outcome 64
Time Frame: From Day 1 to Day 90
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 50 | 22
Days | 1.1 (1.6) | 1.0 (1.9)

79. Secondary Outcome: Difference in Duration Between Longest and Shortest Spotting-only Episodes in Reference Period 2
Description: Reference Period 2 is defined as Day 91 to Day 180 during study treatment.
Time Frame: From Day 91 to Day 180
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 33 | 16
Days | 1.3 (2.0) | 0.8 (1.7)

80. Secondary Outcome: Percentage of Participants With / Without Withdrawal Bleeding at Cycle 1
Description: Withdrawal bleeding is bleeding that occurs when using oral contraceptives (OCs) caused by falling levels and/or taking away external source of estrogen and progestogen toward cycle end
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 101 | 107
Percentage of participants
  without withdrawal bleeding | 24.8 | 2.8
  with withdrawal bleeding | 75.2 | 97.2

81. Secondary Outcome: Percentage of Participants With / Without Withdrawal Bleeding at Cycle 3
Description: as for outcome 80
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 96 | 99
Percentage of participants
  without withdrawal bleeding | 13.5 | 0.0
  with withdrawal bleeding | 86.5 | 100.0

82. Secondary Outcome: Percentage of Participants With / Without Withdrawal Bleeding at Cycle 6
Description: as for outcome 80
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 74 | 75
Percentage of participants
  without withdrawal bleeding | 51.4 | 8.0
  with withdrawal bleeding | 48.6 | 92.0

83. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 1
Description: as for outcome 80
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 76 | 104
Days | 4.3 (2.4) | 4.6 (1.9)

84. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 3
Description: as for outcome 80
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 83 | 99
Days | 4.3 (2.6) | 4.4 (1.5)

85. Secondary Outcome: Length of Withdrawal Bleeding Episodes at Cycle 6
Description: as for outcome 80
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 36 | 69
Days | 3.4 (1.4) | 4.0 (1.3)

86. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 1
Description: Intensity was rated as 1=spotting; 2=light; 3=normal or 4=heavy.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 76 | 104
Scores on a scale | 3.1 (0.8) | 3.7 (0.8)

87. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 3
Description: Intensity was rated as 1=spotting; 2=light; 3=normal or 4=heavy.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 83 | 99
Scores on a scale | 3.2 (0.8) | 3.8 (0.7)

88. Secondary Outcome: Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 6
Description: Intensity was rated as 1=spotting; 2=light; 3=normal or 4=heavy.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 36 | 69
Scores on a scale | 3.0 (1.0) | 3.6 (0.9)

89. Secondary Outcome: Percentage of Participants by Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 1
Description: Withdrawal bleeding is bleeding that occurs when using oral contraceptives (OCs) caused by falling levels and/or taking away external source of estrogen and progestogen toward cycle end. Intensity rated on 4-point scale from 1=spotting to 4=heavy.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 76 | 104
Percentage of participants
  spotting | 22.4 | 7.7
  light | 44.7 | 25.0
  normal | 30.3 | 53.8
  heavy | 2.6 | 13.5

90. Secondary Outcome: Percentage of Participants by Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 3
Description: as for outcome 89
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 83 | 99
Percentage of participants
  spotting | 26.5 | 4.0
  light | 33.7 | 25.3
  normal | 37.3 | 61.6
  heavy | 2.4 | 9.1

91. Secondary Outcome: Percentage of Participants by Maximum Intensity of Withdrawal Bleeding Episodes at Cycle 6
Description: as for outcome 89
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 36 | 69
Percentage of participants
  spotting | 38.9 | 13.0
  light | 27.8 | 26.1
  normal | 27.8 | 47.8
  heavy | 5.6 | 13.0

92. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 1
Description: Onset of withdrawal bleeding was calculated from the end of the exposure to the progestogen component (Day 24 for EV/DNG and Day 21 for EE/LNG). Therefore the count for the onset started at each Cycle on Day 25 for EV/DNG and Day 22 for EE/LNG.
Time Frame: From Day 24 for EV/DNG and Day 21 for EE/LNG to Day 28 for Cycle 1
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 76 | 104
Days | 3.5 (5.0) | 3.4 (2.3)

93. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 3
Description: as for outcome 92
Time Frame: From Day 24 for EV/DNG and Day 21 for EE/LNG to Day 28 for Cycle 3
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 83 | 99
Days | 4.2 (6.5) | 3.6 (2.6)

94. Secondary Outcome: Onset of Withdrawal Bleeding Episodes at Cycle 6
Description: as for outcome 92
Time Frame: From Day 24 for EV/DNG and Day 21 for EE/LNG to Day 28 for Cycle 6
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 36 | 69
Days | 1.1 (1.7) | 3.3 (1.1)

95. Secondary Outcome: Percentage of Participants With Presence or Absence of Intracyclic Bleeding at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 101 | 107
Percentage of participants
  with absence of intracyclic bleeding | 84.2 | 95.3
  with presence of intracyclic bleeding | 15.8 | 4.7

96. Secondary Outcome: Percentage of Participants With Presence or Absence of Intracyclic Bleeding at Cycle 3
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 96 | 99
Percentage of participants
  with absence of intracyclic bleeding | 82.3 | 96.0
  with presence of intracyclic bleeding | 17.7 | 4.0

97. Secondary Outcome: Percentage of Participants With Presence or Absence of Intracyclic Bleeding at Cycle 6
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 74 | 75
Percentage of participants
  with absence of intracyclic bleeding | 83.8 | 94.7
  with presence of intracyclic bleeding | 16.2 | 5.3

98. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 101 | 107
episodes | 0.2 (0.5) | 0.1 (0.3)

99. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 3
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 96 | 99
episodes | 0.2 (0.4) | 0.1 (0.3)

100. Secondary Outcome: Number of Intracyclic Bleeding Episodes at Cycle 6
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 74 | 75
episodes | 0.2 (0.4) | 0.1 (0.3)

101. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 16 | 5
Days | 3.5 (3.4) | 2.4 (1.9)

102. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 3
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 17 | 4
Days | 5.0 (5.2) | 2.8 (2.4)

103. Secondary Outcome: Maximum Length of Intracyclic Bleeding Episodes at Cycle 6
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 12 | 4
Days | 3.5 (1.4) | 5.0 (5.7)

104. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 101 | 107
Days | 0.6 (1.9) | 0.1 (0.8)

105. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 3
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 96 | 99
Days | 0.9 (2.9) | 0.1 (0.7)

106. Secondary Outcome: Number of Intracyclic Bleeding Days at Cycle 6
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 74 | 75
Days | 0.6 (1.4) | 0.3 (1.6)

107. Secondary Outcome: Percentage of Participants by Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 1
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens. Intensity rated on 4-point scale where 1=spotting; 2=light; 3=normal; and 4=heavy.
Time Frame: At Cycle 1 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 16 | 5
Percentage of participants
  spotting | 75.0 | 80.0
  light | 6.3 | 20.0
  normal | 12.5 | 0.0
  heavy | 6.3 | 0.0

108. Secondary Outcome: Percentage of Participants by Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 3
Description: as for outcome 107
Time Frame: At Cycle 3 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 17 | 4
Percentage of participants
  spotting | 64.7 | 75.0
  light | 23.5 | 25.0
  normal | 11.8 | 0.0
  heavy | 0.0 | 0.0

109. Secondary Outcome: Percentage of Participants by Maximum Intensity of Intracyclic Bleeding Episodes at Cycle 6
Description: as for outcome 107
Time Frame: At Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 12 | 4
Percentage of participants
  spotting | 66.7 | 100.0
  light | 8.3 | 0.0
  normal | 16.7 | 0.0
  heavy | 8.3 | 0.0

110. Secondary Outcome: Percentage of Participants With at Least 1 Intracyclic Bleeding Episode
Description: Intracyclic bleeding is any unexpected bleeding episode occurring in cyclical treatment regimens.
Time Frame: Up to Cycle 6 (28 days per Cycle)
Population: All participants in FAS with assessment for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Number analyzed (Participants) | 103 | 107
Percentage of participants
  no | 63.1 | 87.9
  yes | 36.9 | 12.1

ADVERSE EVENTS:
Arm/Group | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) | EE/LNG (Microgynon) + Placebo
Serious Adverse Events (participants affected / at risk) | 3/106 | 0/107
Other Adverse Events (participants affected / at risk) | 32/106 | 11/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) (N=106) | EE/LNG (Microgynon) + Placebo (N=107)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EV/DNG (Natazia, Qlaira, BAY86-5027, SH T00658ID) (N=106) | EE/LNG (Microgynon) + Placebo (N=107)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Influenza (Infections and infestations) | 5 (5) | 2 (2)
Pharyngitis (Infections and infestations) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 9 (31) | 5 (10)
Migraine (Nervous system disorders) | 3 (3) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution must ensure Discloser gives 40 days notice of proposed Publication to Sponsor who may within 40-day period: provide comments, Institution must consider such comments but is not bound to follow them; request delay of Publication for 120 days to allow Sponsor to file patent applications or take other measures to preserve its proprietary rights, Institution must abide by request; request Discloser remove specified Confidential Information, Institution must remove such Information.